CLINICAL TRIAL: NCT03327610
Title: Selecting the Best Ventilator Hyperinflation Settings Based on Physiologic Markers: Randomized Controlled Study
Brief Title: Selecting the Best Ventilator Hyperinflation Settings
Acronym: VHI1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Fernando Silva Guimaraes, Associate Professor, Centro Universitário Augusto Motta
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: VHI1
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Failure; Respiration Disorders
Keywords: Respiratory Therapy; Positive Pressure Respiration; Physical Therapy Modalities
MeSH Terms: conditions — Respiratory Insufficiency; Respiration Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- BASELINE (No Intervention): The subjects were kept in their current ventilatory mode.
- VC-CMV20 (Experimental): Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV) with an inspiratory flow of 20Lpm.
  Interventions: Other: VC-CMV20
- VC-CMV50 (Experimental): Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV) with an inspiratory flow of 50Lpm.
  Interventions: Other: VC-CMV50
- PC-CMV1 (Experimental): Application of a ventilator hyperinflation intervention with Pressure Control Continuous Mandatory Ventilation (PC-CMV1) with an inspiratory time of 1 second.
  Interventions: Other: PC-CMV1
- PC-CMV3 (Experimental): Application of a ventilator hyperinflation intervention with Pressure Control Continuous Mandatory Ventilation (PC-CMV1) with an inspiratory time of 3 seconds.
  Interventions: Other: PC-CMV3
- PSV10 (Experimental): Application of a ventilator hyperinflation intervention with Pressure Support Ventilation (PSV) with a cycling off of 10% of peak inspiratory flow.
  Interventions: Other: PSV10
- PSV25 (Experimental): Application of a ventilator hyperinflation intervention with Pressure Support Ventilation (PSV) with a cycling off of 25% of peak inspiratory flow.
  Interventions: Other: PSV25

INTERVENTIONS:
Other: VC-CMV20 — Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV). The inspiratory flow was set at 20Lpm and the tidal volume was increased in steps of 200mL until the peak airway pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: VC-CMV20
Other: VC-CMV50 — Application of a ventilator hyperinflation intervention with Volume Control Continuous Mandatory Ventilation (VC-CMV). The inspiratory flow was set at 50Lpm and the tidal volume was increased in steps of 200mL until the peak airway pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: VC-CMV50
Other: PC-CMV1 — Application of a ventilator hyperinflation intervention with Pressure Control Continuous Mandatory Ventilation (PC-CMV1). The inspiratory time was set at 1 second and the pressure control was increased until a peak pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: PC-CMV1
Other: PC-CMV3 — Application of a ventilator hyperinflation intervention with Pressure Control Continuous Mandatory Ventilation (PC-CMV1). The inspiratory time was set at 3 seconds and the pressure control was increased until a peak pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: PC-CMV3
Other: PSV10 — Application of a ventilator hyperinflation intervention with Pressure Support Ventilation (PSV). The cycling off was set at 10% of peak inspiratory flow and the pressure support was increased until a peak pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: PSV10
Other: PSV25 — Application of a ventilator hyperinflation intervention with Pressure Support Ventilation (PSV). The cycling off was set at 25% of peak inspiratory flow and the pressure support was increased until a peak pressure of 40cmH2O was achieved. After achieving the target pressure, this ventilatory regimen lasted 15 minutes. Positive end expiratory pressure and the inspired oxygen fraction were not modified.
  Arms: PSV25

SUMMARY:
Ventilator hyperinflation (VHI) has been shown to be effective in improving respiratory mechanics, secretion removal, and gas exchange in mechanically ventilated patients; however, there are no recommendations on the best ventilator settings to perform the technique. Thus, the aim of this study was to compare six modes of VHI, concerning physiological markers of efficacy and safety criteria, in order to support the optimal VHI settings selection for mechanically ventilated patients. In a randomized, controlled and crossover study, 30 mechanically ventilated patients underwent 6 modes of ventilator hyperinflation. The maximum expansion (tidal volume), expiratory flow bias criteria (inspiratory and expiratory flow patterns), overdistension (alveolar pressure), asynchronies and hemodynamic variables (mean arterial pressure and heart rate) were assessed during the interventions.

DETAILED DESCRIPTION:
Background: Ventilator Hyperinflation (VHI) has been shown to be effective in improving respiratory mechanics, secretion removal, and gas exchange in mechanically ventilated patients; however, there are no recommendations on the best ventilator settings to perform the technique. Thus, the aim of this study was to compare six modes of VHI, concerning physiological markers of efficacy and safety criteria, in order to support the optimal VHI settings selection for mechanically ventilated patients.

Methods: In a crossover study, every included mechanically ventilated patient underwent six modes of VHI in a randomized order: Volume Control Continuous Mandatory Ventilation (VC-CMV) with inspiratory flow = 20Lpm (VC-CMV20), VC-CMV with inspiratory flow = 50Lpm (VC-CMV50), Pressure Control Continuous Mandatory Ventilation (PC-CMV) with inspiratory time = 1s. (PC-CMV1), PC-CMV with inspiratory time = 3s. (PC-CMV3), Pressure Support Ventilation (PSV) with cycling off = 10% of peak inspiratory flow (PSV10), and PSV with cycling off = 25% of peak inspiratory flow (PSV25). The maximum expansion (tidal volume), expiratory flow bias criteria (inspiratory and expiratory flow patterns), over-distension (alveolar pressure), asynchronies and hemodynamic variables (mean arterial pressure and heart rate) were assessed during the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for more than 48h

Exclusion Criteria:

* mucus hypersecretion (defined as the need for suctioning < 2-h intervals),
* absence of respiratory drive,
* atelectasis,
* severe bronchospasm,
* positive end expiratory pressure > 10cmH2O,
* PaO2-FiO2 relationship < 150,
* mean arterial pressure < 60mmHg,
* inotrope requirement equivalent to >15 ml/h total of adrenaline and noradrenalin,
* intracranial pressure > 20mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Peak inspiratory to expiratory flow ratio | Ten minutes after the onset of intervention.
  Dichotomous variable, defined as achieving a peak inspiratory flow rate (PIFR) less than 90% of the peak expiratory flow rate (PEFR)
Peak expiratory flow higher than 40 Lpm | Ten minutes after the onset of intervention.
  Dichotomous variable, defined as achieving a PEFR higher than 40 l/min
Difference between peak inspiratory and expiratory flows. | Ten minutes after the onset of intervention.
  Dichotomous variable, defined as achieving a difference higher than 17Lpm.
Pulmonary expansion | Ten minutes after the onset of intervention.
  Percentage of tidal volume above the normal tidal volume (estimated as 6mL/kg).

SECONDARY OUTCOMES:
Mean arterial pressure | Ten minutes after the onset of intervention.
  Mean arterial pressure verified using the multi-parameter monitor.
Heart Rate | Ten minutes after the onset of intervention.
  Heart rate verified using the multi-parameter monitor.

CONTACTS AND LOCATIONS:
Overall Officials: FERNANDO S GUIMARAES, PhD, Study Chair — Centro Universitário Augusto Motta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berney S, Denehy L. A comparison of the effects of manual and ventilator hyperinflation on static lung compliance and sputum production in intubated and ventilated intensive care patients. Physiother Res Int. 2002;7(2):100-8. doi: 10.1002/pri.246. PMID 12109234
- [Background] Lemes DA, Zin WA, Guimaraes FS. Hyperinflation using pressure support ventilation improves secretion clearance and respiratory mechanics in ventilated patients with pulmonary infection: a randomised crossover trial. Aust J Physiother. 2009;55(4):249-54. doi: 10.1016/s0004-9514(09)70004-2. PMID 19929767
- [Background] Thomas PJ. The effect of mechanical ventilator settings during ventilator hyperinflation techniques: a bench-top analysis. Anaesth Intensive Care. 2015 Jan;43(1):81-7. doi: 10.1177/0310057X1504300112. PMID 25579293
- [Background] Ntoumenopoulos G, Shannon H, Main E. Do commonly used ventilator settings for mechanically ventilated adults have the potential to embed secretions or promote clearance? Respir Care. 2011 Dec;56(12):1887-92. doi: 10.4187/respcare.01229. Epub 2011 Jun 17. PMID 21682986
- [Background] Anderson A, Alexanders J, Sinani C, Hayes S, Fogarty M. Effects of ventilator vs manual hyperinflation in adults receiving mechanical ventilation: a systematic review of randomised clinical trials. Physiotherapy. 2015 Jun;101(2):103-10. doi: 10.1016/j.physio.2014.07.006. Epub 2014 Oct 6. PMID 25453540
- [Background] Davies JD, Senussi MH, Mireles-Cabodevila E. Should A Tidal Volume of 6 mL/kg Be Used in All Patients? Respir Care. 2016 Jun;61(6):774-90. doi: 10.4187/respcare.04651. PMID 27235313
- [Background] de Wit M. Monitoring of patient-ventilator interaction at the bedside. Respir Care. 2011 Jan;56(1):61-72. doi: 10.4187/respcare.01077. PMID 21235839
- See also: Researchgate profile (Chair researcher) — https://www.researchgate.net/profile/FERNANDO_GUIMARAES
- See also: ResearcherID profile (Chair researcher) — http://www.researcherid.com/ProfileView.action?returnCode=ROUTER.Unauthorized&Init=Yes&SrcApp=CR&queryString=KG0UuZjN5WkrS6qTMqySbml%252FKME%252FypfZgkjPia93VtU%253D